CLINICAL TRIAL: NCT04193605
Title: Feasibility of the Mindfulness-Based Stress Reduction Intervention for Black Women Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Crystal C. Lambert, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K23AT010567 (NIH); K23AT010567 (NIH)
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: HIV Infections; Health Behavior
MeSH Terms: conditions — HIV Infections; Health Behavior | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Stress Reduction (Active Comparator): MBSR sessions received by the treatment group will include an orientation, approximately 8 intervention sessions, and an exit interview.
  Interventions: Behavioral: Mindfulness
- Standard of Care (No Intervention): The control condition will continue receiving usual care or standard of care.

INTERVENTIONS:
Behavioral: Mindfulness — The traditional MBSR intervention consists of the following: (1) a series of eight weekly session of 2.5 to 3 hours; (2) a silent retreat during the sixth week; (3) daily home assignments including formal and informal mindfulness practices; and (4) didactic presentations on stress and the consequences of stress. We are culturally tailoring the intervention with the goal of maintain fidelity.
  Arms: Mindfulness Based Stress Reduction

SUMMARY:
The investigator propose to culturally adapt the mindfulness-based stress reduction (MSBR) intervention for Black/African American women living with HIV (WLWH) to reduce stress and enhance HIV self-care behaviors and viral load (VL) suppression, which has the potential to attenuate prominent racial and gender disparities experienced by Black WLWH in the US. Specifically, the investigator aims to 1) culturally adapt the MBSR intervention for Black WLWH using ADAPT-ITT; 2) pre-pilot the adapted intervention via an open non-randomized pilot study to further refine the culturally adapted intervention; and 3) conduct a 2-armed randomized pilot test of the behavioral intervention compared to standard of care to assess the feasibility and acceptability the adapted MBSR intervention for Black WLWH. The investigator hypothesis that the adapted intervention will be feasible and acceptable to member of the target population.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender females
* HIV seropositive
* 18 years of age or older
* English speaking
* An active patient at the local HIV ambulatory clinic in Alabama.

Exclusion Criteria:

* Non-English speaking
* Appear temporarily impaired (e.g., intoxicated)
* Not willing to or legally unable to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants are required to be born a female.
Enrollment: 48 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UAB School of Nursing, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
UAB maintains the following universal data sharing policy for all investigators:
  1. Data will be made available, in accordance with the NIH Data Sharing Policy (http://grants.nih.gov/grants/policy/data_sharing) to all researchers in both the private and public sector free or for a nominal charge and with minimal restriction. In some cases the institution may determine that the public and the research community are better served by a licensing program whether or not patents have been filed. This may be relevant, for example, if a tool is best distributed under license to guarantee reagent availability and quality.
  2. As a means of sharing knowledge, NIH encourages grantees to arrange for publication of NIH-supported original research in primary scientific journals. We therefore will strive to publish our findings in a timely manner and acknowledge that the research was supported by the NIH.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness Based Stress Reduction | Standard of Care
Started | 24 | 24
Completed | 21 | 20
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Based Stress Reduction | Standard of Care | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (10.9) | 47.4 (7.5) | 47.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 24 | 48
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Intervention Measure
Description: Feasibility was measured using a four-item feasibility of intervention measure. Each item is scored using a Likert-like scale ranging from "1" completely disagree to "5" completely agree. Higher scores indicate greater feasibility. The minimum total score is 4 points, and the maximum total score is 20.
Time Frame: Immediately after the intervention(which consists of an orientation followed by eight weekly sessions, consistent with MSBR interventions), the measure was collected within one week of completing the final session.
Population: Participants in the standard of care did not receive the intervention. Therefore, data was not collected or analyzed on these participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Based Stress Reduction | Standard of Care
Number analyzed (Participants) | 21 | 0
units on a scale | 18 (2.4) |

ADVERSE EVENTS:
Time Frame: The intervention was eight weeks long. Therefore, adverse events were collected for 8 weeks.
Arm/Group | Mindfulness Based Stress Reduction | Standard of Care
All-Cause Mortality (participants affected / at risk) | 1/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

LIMITATIONS AND CAVEATS:
This is a feasibility. Therefore, we were not powered to detect changes in specific outcome measures. The primary outcome was feasibility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-31): https://cdn.clinicaltrials.gov/large-docs/05/NCT04193605/Prot_SAP_000.pdf